CLINICAL TRIAL: NCT05734729
Title: Clinical Validation of Programmable Chest and Abdominal Drain Fluid Regulator to Reduce Morbidity, Care Requirements, and Improve Outcomes: First-In-Human Medical Device Study
Brief Title: Clinical Validation of Programmable Drain Fluid Regulator to Reduce Morbidity, Care Requirements, and Improve Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Jessica Quah Li Shan, Consultant, Changi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFFIDRAIN
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Pleural Effusion; Ascites
Keywords: Medical device; Pleural effusion; Ascites; Drainage; Novel
MeSH Terms: conditions — Pleural Effusion; Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pleural Arm (Experimental): Patient's maximum volume is 1 litre per hour, not to exceed total 4 litres over 4 hours
  Interventions: Device: EFFIDRAIN; Device: Manual drainage system
- Ascites arm (Experimental): Patient's maximum volume is 3 litre per hour, not to exceed total 15 litres over 5 hours
  Interventions: Device: EFFIDRAIN; Device: Manual drainage system

INTERVENTIONS:
Device: EFFIDRAIN — . Effidrain is a progammable, light-weight, portable drain regulator that can control the rate and volume of body fluid being drained, while empowering the user with information on dynamic changes of pressure within the body cavity being drainged. It is able to adapt to existing drainage systems via a standard medical luer taper connector, and comes with a failsafe system to alert users of drainage irregularities.
Device: Manual drainage system — drainage systems required manual control and are unautomated; consequent unintended rapid intravascular and extravascular fluid shifts may result in clinical instability.

SUMMARY:
The goal of this Effidrain first-in-human medical device trial is to improve the outcomes of patients with pleural effusions and ascites.

The main aims are:

* The primary aim of this first-in-man device pivotal study (n=120) is to demonstrate that the body fluid drain regulator can perform the function of pleural or ascites drainage, accurately and precisely.
* The secondary aims are related to explore the effects of Effidrain on health-related outcomes:

  1. The investigators hypothesize that Effidrain can reduce the time that the subject requires a pleural or abdominal drain in-situ, compared to conventional care.
  2. The investigators hypothesize that the time required for healthcare workers to perform post-procedure monitoring for subjects that require pleural or abdominal drainage using Effidrain, would be reduced compared to conventional care. The effect of technology on physician and nursing hours required for drain care, and cost-effectiveness of the intervention will be studied

Participants will be randomized to control and intervention group. Control group will be receiving treatment using manual drainage system while intervention group will be using Effidrain machine.

Participants and Nurses from both control and intervention group will be asked to fill participant/nurses questionnaire form respectively.

DETAILED DESCRIPTION:
The mission of the Effidrain first-in-human medical device trial is to improve the outcomes of patients with pleural effusions and ascites.

The primary aim of this first-in-man device pivotal study (n=120) is to demonstrate that the body fluid drain regulator can perform the function of pleural or ascites drainage, accurately and precisely.

The primary hypothesis is that the group of patients with device drainage intervention would be able to demonstrate actual fluid drainage not more than 110% of the physician-prescribed drainage volume and time.

The secondary aims are related to explore the effects of Effidrain on health-related outcomes:

1. The investigators hypothesize that Effidrain can reduce the time that the subject requires a pleural or abdominal drain in-situ, compared to conventional care.
2. The investigators hypothesize that the time required for healthcare workers to perform post-procedure monitoring for subjects that require pleural or abdominal drainage using Effidrain, would be reduced compared to conventional care. The effect of technology on physician and nursing hours required for drain care, and cost-effectiveness of the intervention will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Pleural effusion or ascites as the primary indication for chest or abdominal drain insertion
* Expected ascites drainage volume more than 1 Litre or at least moderate sized pleural effusion (occupying more than one-third hemi-thorax)
* uncomplicated chest or abdominal drain insertion
* Adults aged 21 years, able to provide (or surrogate able to provide) consent.

Exclusion Criteria:

* Vulnerable persons, including but not limited to, pregnant women and prisoners
* Hemodynamic instability, defined by heart rate more than 120 beats per minutes and blood pressure less than systolic 90mmHg
* Haemothorax or Haemoperitoneum
* pneumothorax or pneumoperitoneum
* chest or abdominal drain insertion => 48 hours with more than estimated 50% of total body cavity fluid drained

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
demonstrate that the Effidrain can perform the function of pleural and ascites drainage in human subjects accurately and precisely | after 72 hours of usage per patient
  A session completed by the medical device not exceeding 10% volume of the physican precribed drainage volume is considered a success and scored as completely meeting device efficacy criteria.
  A session completed by the medical device not exceeding 25% volume of the physican precribed drainage volume is considered a success and scored as partially meeting device efficacy criteria.
  A session completed by the medical device exceeding 25% volume of the physican precribed drainage volume is considered a failure and scored as not meeting device efficacy criteria.

SECONDARY OUTCOMES:
Reduction in time that a subject requires a chest or abdominal drain in-situ | Total of 4 hours for Pleural arm and 5 hours for Ascites arm
  Mean difference between of physician-planned drainage volume and time required, vs actual drainage volume and time, in both intervention and control arms will be analysed using T-tests.
Reduction in time required for post-procedure monitoring by healthcare workers | after 72 hours of usage per patient
  Further analysis involve quantifying the effect of Effidrain on health-related outcomes such as:
  1. Reduction in time that a subject requires a chest or abdominal drain in-situ
  2. Reduction in time required for post-procedure monitoring by healthcare workers
  3. Inpatient hospitalisation days The median times for the variables above would be compared between interventional and control groups using Mann Whitney U tests
Improvement in cost-effectiveness of care for each inpatient episode of pleural effusion or ascites that requires drainage. | after 72 hours of usage per patient
  To estimate the costs, the following cost and probabilities data will be extracted from the different databases, including the hospital's electronic database:
  1. Number of patients requiring pleural and abdominal drainage in Changi General Hospital per year
  2. Costs of developing the Effidrain from hospital perspective
  3. Costs of maintaining the Effidrain from hospital perspective (including man-hours and actual expenditure incurred by the hospital)
  4. Man-hours and unit cost of man-hours in conducting pleural and abdominal drainage using the Effidrain
  5. Man-hours and unit cost of man-hours in conducting pleural and abdominal drainage using manual drainage
  6. Length of stay of patients using the Effidrain and the manual drainage

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore